CLINICAL TRIAL: NCT00446758
Title: Trial of Zinc and HIV Progression in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Thrasher Research Fund (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Eduardo Villamor, Adjunct Associate Professor of International Nutrition, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14511
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: Zinc; HIV; Infants; Children; Morbidity; Child health outcomes; treatment naive; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc (Experimental): zinc (as zinc sulphate) 12.5 mg orally per day (6.25 mg in children < 12 mo)
  Interventions: Dietary Supplement: Zinc
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — zinc effervescent tablets: 6.25mg to infants ≤12 months and 12.5 mg to children > 12 months.

SUMMARY:
To examine whether daily oral zinc supplementation to HIV-infected Tanzanian preschool children reduces diarrheal and respiratory morbidity, delays HIV disease progression, and improves growth.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether daily oral zinc supplementation to HIV-infected Tanzanian preschool children reduces diarrheal and respiratory morbidity, delays HIV disease progression, and improves growth.

ELIGIBILITY:
Inclusion Criteria:

* HIV Infected Children under 60 months of age presenting at HIV treatment clinics in Dar es Salaam, Tanzania

Exclusion Criteria:

Eligible for ART: CD4 cell counts < 20% or above pediatric clinical stage of HIV disease 3 according to WHO staging system.

Severe acute malnutrition; Major congenital malformations

Ages: 6 Weeks to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 440 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Morbidity from respiratory and diarrheal infections, HIV disease progression | every 4 to 6 months until the end of follow-up

SECONDARY OUTCOMES:
growth in height and weight | every 4 to 6 months until the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Villamor, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimbili University College of Health Sciences, Dar es Salaam, Tanzania